CLINICAL TRIAL: NCT00822705
Title: Inhibition of Food Intake in Response to Oral GLP-1 and Peptide YY3-36: a Phase 1 Study
Brief Title: Inhibition of Food Intake in Response to Oral GLP-1 and Peptide YY3-36
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Prof. Christoph Beglinger, University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EKBB 127/07; SNF grant 320000-118330
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Anti Obesity Agent
Keywords: Appetite, energy consumption, gastrointestinal hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ORAL GLP-1, TABLET (Active Comparator)
  Interventions: Drug: Placebo tablet
- Oral PYY3-36 (Active Comparator)
  Interventions: Drug: Placebo tablet
- Oral GLP-1 plus oral PYY3-36 (Active Comparator)
  Interventions: Drug: Placebo tablet
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: Placebo tablet — Control arm

SUMMARY:
Interaction of GLP-1 and PYY3-36 in the inhibition of food intake in healthy subjects

DETAILED DESCRIPTION:
PYY3-36 and GLP-1 are two classical gastrointestinal peptides, which are released into the circulation during meals from L-cells of the distal gut; there is compelling evidence that each participates in the control of appetite regulating individual meal sizes in healthy subjects, but also in patients with obesity or diabetes type II. The regulation of human eating habits is, however, highly complex and our understanding of appetite control is far from complete. In many areas our knowledge is rather rudimentary; little is known, to give an example, about the importance of individual signals and their interactions.

From studies in animals and humans it is known that individual satiety signals can interact: contributions of glucagon and CCK produced functionally synergistic inhibitions of feeding in rats, that is, simultaneous injection of the two peptides inhibited feeding significantly more than the sum of their individual effects. In contrast, we have been unable to show in healthy volunteers any interaction between GLP-1 and CCK33; the simultaneous infusion of CCK33 and GLP-1 resulted in an infra-additive reduction in meal size, which led us to suggest that the two peptides could even interact antagonistically.

To further explore potential interactions between these two well-known satiety signals, we plan to investigate the effects of individual doses of PYY3-36 and GLP-1, and their interaction in the control of food intake and satiety in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects
* no evidence of disease
* no history of gastrointestinal or endocrine disorders

Exclusion Criteria:

* alcohol and drug abuse
* history of gastrointestinal or endocrine disorders
* female subjects

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Energy consumption | 1 hour food consumption

SECONDARY OUTCOMES:
Appetite feelings, plasma kinetics adverse events | adeverse events during study (3 months)

CONTACTS AND LOCATIONS:
Overall Officials: CHRISTOPH BEGLINGER, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Clinical Research Center, University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Steinert RE, Poller B, Castelli MC, Drewe J, Beglinger C. Oral administration of glucagon-like peptide 1 or peptide YY 3-36 affects food intake in healthy male subjects. Am J Clin Nutr. 2010 Oct;92(4):810-7. doi: 10.3945/ajcn.2010.29663. Epub 2010 Aug 18. PMID 20720259